CLINICAL TRIAL: NCT04048915
Title: 3Hs Family Drama Project (Phase 2)
Brief Title: Family Drama Project II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Boys' and Girls' Clubs Association of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 15-464
Record Dates: First submitted 2019-07-29; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Family Health, Happiness and Harmony; Physical Health
Keywords: Family well-being; Healthy Eating; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Long live drama (Experimental): Primary school students watched an interactive long live drama (90 minutes) in schools. DVD and worksheets were also distributed to students and asked them to watch the DVD and finish the worksheets with their parents.
  Interventions: Behavioral: Long live drama
- Short live drama (Experimental): Primary school students watched an interactive short live drama (60 minutes) in schools. DVD and worksheets were also distributed to students and asked them to watch the DVD and finish the worksheets with their parents.
  Interventions: Behavioral: Short live drama
- Waitlist control (No Intervention): Primary school students received no intervention during the 3-month study period. After the study finished, the students watched either short or long live drama, and DVD with worksheets were distributed to students and they were invited to share with their parents.

INTERVENTIONS:
Behavioral: Long live drama — The interactive live 90-minute drama and DVD conveyed educational information on healthy living habits (including physical activity and healthy eating) as well as the importance and suggested methods to enhance family well-being. Students were encouraged to share the information on healthy living habits and watched the DVD with their parents.
  Worksheets were given to all students and encouraged to finish the worksheets with their parents.
  Arms: Long live drama
Behavioral: Short live drama — The interactive live 60-minute drama and DVD conveyed educational information on healthy living habits (including physical activity and healthy eating) as well as the importance and suggested methods to enhance family well-being. Students were encouraged to share the information on healthy living habits and watched the DVD with their parents.
  Worksheets were given to all students and encouraged to finish the worksheets with their parents.
  Arms: Short live drama

SUMMARY:
A harmonious family relationship has significant effects on the psychological well-being and development of children. Good communication between parents and children is a crucial element for family health, happiness and harmony. However, communication within Hong Kong families is vastly inadequate partly due to our busy urban lifestyle.

The 3Hs Family Drama Project (Phase 2) was an enhanced version of the 3Hs Family Drama Project to promote health, happiness, harmony (3Hs), healthy eating and physical activity in primary school students. Students watched the interactive live drama (long or short version) and are given DVD and worksheets. Students were encouraged to watch the DVD with other family members at home. The present study aimed to evaluate the effectiveness and satisfaction levels of teachers, parents and students towards the drama project.

DETAILED DESCRIPTION:
3Hs Family Drama Project (Phase 2) was an intervention to enhance the 3Hs through increasing interaction and communication between parents and children. Healthy eating and physical activity were also promoted. The drama project conducted 100 drama performances (either in the long or short version) in primary schools during the 2015-16 school year. The main targets were Primary 3 to 5 (P3-5) students and their families. Students would take home a DVD of the drama to watch and worksheets to complete with parents and other family members.

The goals of the study were to evaluate the effectiveness of the project to enhance health, happiness, harmony (3Hs), healthy eating and physical activity and participants' satisfaction levels towards the drama project.

Quantitative assessments were used to evaluate the effectiveness of the project. Process evaluations were performed in randomly selected students, parents and teachers to evaluate the process of each component of the program. Qualitative and quantitative assessments were used. Students, parents and teachers were asked to express their views on a questionnaire. Feedback from students was also collected through small group discussions, while that of parents was collected through telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

Students: (both the Intervention group and waitlist control group)

* 1. Students who can read Chinese.
* 2. Primary 3 to 5 students in participating primary schools.

Parents: (Intervention group only)

* 1. Parents who can read Chinese.
* 2. With at least one primary school child.

School teachers: (Intervention group only)

* 1. Teachers who can read Chinese.

Exclusion Criteria:

* Students, parents or teachers who cannot read Chinese.

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7026 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change in family health, happiness and harmony (3Hs) | baseline and 3 months
  Health, happiness and harmony (3Hs) were assessed by family well-being scale. Perceived family harmony and health were measured by 2 questions on a scale ranging from 1 to 5, whereas perceived family happiness was measured by a single question on a scale ranging from 1 to 4. The higher score the better.

SECONDARY OUTCOMES:
Change in parent-child interactions | baseline, 1 month and 3 months
  Students were asked whether they performed the 12 mentioned activities (e.g. watching movies with parents) in the past 7 days.
Change in knowledge on healthy eating | baseline, 1 month and 3 months
  Students were asked by 4 questions: 1)Do typical photo chips contain salt; 2)Will drinking sugary drinks affect weight; 3)Will more sedentary behaviours affect weight and 4)How many cubes of sugar are in a can of coke. The former 3 questions were given with 4 options, while the latter was given with 8 options. Each corrected answer scores 1 and a sum of scores from the 4 questions were deemed a measurement of knowledge.
Change in behavior on physical activity | baseline, 1 month and 3 months
  Students were asked to report the number of days (0-7) of simple exercise and at least 60 minutes moderate-to-vigorous physical activity in the past 7 days.
Satisfaction towards the live drama, song and interactive parts | Immediately after the live drama
  Students were asked to rate the live drama, song and interactive parts on a scale ranging from 1 to 5 scale and the lower score the more satisfied.
Change in family health, happiness and harmony (3Hs) | baseline and 1 month
  Health, happiness and harmony (3Hs) were assessed by family well-being scale. Perceived family harmony and health were measured by 2 questions on a scale ranging from 1 to 5, whereas perceived family happiness was measured by a single question on a scale ranging from 1 to 4. The higher score the better.
Changes in body mass index | baseline and 1 month
  Body mass index was calculated from the measured weight and height
Changes in physical fitness (muscle strength) | baseline and 1 month
  Muscle strength was assessed through a dynamometer
Changes in physical fitness (muscle endurance) | baseline and 1 month
  Muscle endurance of legs was assessed through a simple fitness test "Squat".
Changes in physical fitness (muscle endurance) | baseline and 1 month
  Muscle endurance was assessed through a simple fitness test "Plank".
Change in fruit and vegetable consumption | baseline, 1 month and 3 months
  Students were asked to report the number of days (0-7) of consuming at least 2 servings of fruit and 3 servings of vegetables in the past 7 days.
Satisfaction towards the DVD and worksheets | 1 month
  Students were asked to rate the DVD and worksheets on a scale ranging from 1 to 5 and the lower score the more satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Yin Ho, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Local primary schools, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No